CLINICAL TRIAL: NCT05689489
Title: Use of Puzzle Method in Psychiatric Nursing Teaching: A Randomized Controlled Study
Brief Title: Use of Puzzle Method in Psychiatric Nursing Teaching
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Emel Erdeniz Güreş, Research Assistant, Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 0000-0003-3949-2770
Record Dates: First submitted 2023-01-09; First posted 2023-01-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Psychiatric Nursing
Keywords: Education; Puzzle; Psychiatric Nursing

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Puzzle (Experimental)
  Interventions: Other: Puzzle Method
- control group (Active Comparator)
  Interventions: Other: Ongoing Education

INTERVENTIONS:
Other: Puzzle Method — While preparing the puzzle to be used in the study, the puzzle preparation program will be used (Crossword Puzzle Maker). Students in the initiative group will be asked to solve a total of 6 puzzles, one puzzle each week. The answers to the prepared puzzles will cover the theoretical course topics of psychiatric nursing. In the puzzles, students will be expected to place their answers in the specified rows and columns. Students will be asked to solve puzzles individually. In addition, the answer to each puzzle will be found on the reverse on the back page. Students will be reminded that there is no time limit for solving the puzzles. Researchers will guide students while students solve puzzles.
  Arms: Puzzle
Other: Ongoing Education — Students in the control group will only take the theoretical course of psychiatric nursing.
  Arms: control group

SUMMARY:
Objective: It is thought that the puzzle technique and teaching method will be useful in teaching psychiatric nursing in order to facilitate the learning of psychiatric symptoms and findings and to increase awareness in mental state examination. For this reason, the research was planned to examine the effectiveness of the puzzle technique in learning psychiatric symptoms and findings in psychiatric nursing students.

Design: This study was planned in a randomized controlled experimental design.

Method

Place and Time The research is planned to be carried out between November and January 2022 at a foundation university.

Population and Sample of the Research The population of the research will be 108 students enrolled in the nursing program of a foundation university and taking the "Psychiatric Nursing" course in the fall semester of the 2022-2023 academic year.

In the study, it is aimed to reach the entire universe, not selecting the sample. The students in the universe, who accepted to participate in the study and completed the pre-test, will be assigned to the intervention and control groups by randomization with the help of a generator on the www.random.org website by being numbered according to their order in the student list.

Hypothesis: Students who use puzzle method in teaching psychiatric nursing have higher knowledge levels than students who do not.

ELIGIBILITY:
Inclusion Criteria:

* Registered in the nursing department of the university where the research will be conducted,
* Taking a psychiatric nursing course in the fall semester of the 2022-2023 academic year,
* Taking the Psychiatric Nursing course for the first time,
* Does not have a communication problem at a level that prevents the conversation,
* Students who volunteer to participate in the research will be included in the research.

Exclusion Criteria:

* Not registered in the nursing department of the university where the research will be conducted,
* Not taking a psychiatric nursing course in the fall semester of the 2022-2023 academic year,
* Taking the Psychiatric Nursing course for the second time,
* Having a communication problem at a level that prevents the conversation,
* Students who do not volunteer to participate in the research will not be included in the research.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2023-01-09 (Actual)

PRIMARY OUTCOMES:
Descriptive Characteristics Form | 1 week
  Demographic characteristics of students
Information Form for Concepts Used in the Field of Psychiatric Nursing | for 6 weeks
  It is a form consisting of twenty-five items, prepared by the researchers based on the literature, in order to determine the level of knowledge of the students about the concepts used in the field of psychiatric nursing. While fifteen of the items were correct, ten of them were incorrectly stated. In the form, students were asked to mark one of the statements I agree or disagree for each item. Students got 4 points for each correct answer they determined. The lowest score that can be obtained from the form was "0" and the highest score was "100". The content validity index obtained from the experts was found to be 97%.

CONTACTS AND LOCATIONS:
Locations (1):
- Uskdar University, Istanbul, Umraniye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No